CLINICAL TRIAL: NCT05592457
Title: Role of Non-contrast MDCT in the Assessment of Upper Urinary Tract Calculi Post ESWL to Predict Its Success Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Essam, principle investigator, Assiut University
Other Study IDs: MDCT in ESWL
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Urinary Stone
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: MSCT — multislice computed tomography

SUMMARY:
Urinary stones are a common disease affecting one in 11 people . Their clinical presentation varies from being silent to severe loin pain owing to urinary obstruction. Currently, ESWL is the treatment of choice for most renal calculi ⩽30 mm, with success rates of 60-99%. Although many treatment options exist, ESWL has the advantages of simplicity and non-invasiveness. In contrast, failure of a first ESWL attempt requires a follow-up ESWL procedure, or an alternative procedure, both of which increase medical costs.

Advancements in imaging have significantly contributed to this process. In the mid- 1990s, computed tomography (CT) began to replace intravenous urography (IVU), abdominal films (KUB), and ultrasound (US) in stone diagnosis. Studies demonstrated that CT had superior sensitivity and specificity for stone diagnosis compared to the aforementioned modalities. Now non-contrast multidetector CT (NC-MDCT) is the gold standard for the detection of urinary system calculi. CT is also clinically useful as it can show alternate renal and non-renal pathology if present.

Many factors have been reported to predict ESWL outcome, such as skin-to-stone distance (SSD), stone size, stone location, multiplicity, the energy used, and Hounsfield Unit (HU) values measured by non-contrast computed tomography (NCCT).

DETAILED DESCRIPTION:
Excellent fragmentation results are produced using ESWL. However, the retention of post-ESWL fragments in the kidney continues to be a significant medical issue. Only 32% of calcium stone patients in research were found to remain stone-free for 12 months following ESWL, according to the results. As a result, it appears that fragment growth and persistence are frequent after ESWL [10].

The first ESWL residual that is accessible must undergo a thorough stone analysis to properly carry out the subsequent treatments to prevent relapse or recurrent stone because stone-free rates after ESWL are directly connected to stone placement, size, number, and composition

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years.
* stone size up to 25 mm for renal pelvic stones and up to 15 mm for upper ureteric stones.
* SSD < 11 cm.

Exclusion Criteria:

* any patient with contraindications to ESWL as
* uncontrolled urinary infection.
* clotting alterations.
* aortic or renal artery aneurysm.
* pregnancy.
* serious skeletal malformations.
* serious obesity and or contraindications to CT as pregnancy.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Firstly All studies were performed by using a CT device.
  * the mean Hounsfield unit was calculated. The skin-to-stone distance (SSD) was calculated by measuring three distances from the stone to the skin at 0, 45, and 90°;
  * after the first session of ESWL by one to three weeks Low dose NCCT(MA=175)will be done to determine the measurements of the fragments or the stone if not fragmented including their density and size will be taken, For the density, if decreased or not changed continuation versus stop will be evaluated, while for the size the fragmentation will be assessed as 1- complete fragmentation is the fragment size <4 mm, 2- partial fragmentation if size = 4-5 mm and 3- incomplete fragmentation if the size of fragment more than or equal 6 mm.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
ct follow up during swl | 3 weeks
  Correlation between the stone density before and during ESWL sessions to determine if this predicts the success prevent new ESWL.
stone Hounsfield | 3weeks
  Determine the role of the density of the residual stone fragments in the prediction of the complication during ESWL.

SECONDARY OUTCOMES:
density of stone and other factors | 3weeks
  Correlate between stone density and other factors in the prediction of the success of ESWL.

CONTACTS AND LOCATIONS:
Overall Officials: gehan sayed, MD, Study Director — Assiut University; Doria mohamed, md, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolf JS Jr, Clayman RV. Percutaneous nephrostolithotomy. What is its role in 1997? Urol Clin North Am. 1997 Feb;24(1):43-58. doi: 10.1016/s0094-0143(05)70353-0. PMID 9048851
- [Background] Rassweiler JJ, Renner C, Chaussy C, Thuroff S. Treatment of renal stones by extracorporeal shockwave lithotripsy: an update. Eur Urol. 2001 Feb;39(2):187-99. doi: 10.1159/000052435. PMID 11223679
- [Background] Johnson EK, Faerber GJ, Roberts WW, Wolf JS Jr, Park JM, Bloom DA, Wan J. Are stone protocol computed tomography scans mandatory for children with suspected urinary calculi? Urology. 2011 Sep;78(3):662-6. doi: 10.1016/j.urology.2011.02.062. Epub 2011 Jun 30. PMID 21722946
- [Background] Weld KJ, Montiglio C, Morris MS, Bush AC, Cespedes RD. Shock wave lithotripsy success for renal stones based on patient and stone computed tomography characteristics. Urology. 2007 Dec;70(6):1043-6; discussion 1046-7. doi: 10.1016/j.urology.2007.07.074. PMID 18158009